CLINICAL TRIAL: NCT02613442
Title: Factors Affecting Aqueous Humor Outflow Facility in Patients with Uveitis
Status: Withdrawn | Type: Observational
Why Stopped: Due to uveitis specialist leaving our University
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0749-15-FB
Record Dates: First submitted 2015-11-12; First posted 2015-11-24 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: UVeitis; Glaucoma
MeSH Terms: conditions — Uveitis; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Objective: To determine the clinical variables that influence aqueous outflow facility (Co) and intraocular pressure (IOP) in uveitis.

Uveitic glaucoma is potentially blinding and occurs in 17-46% of chronic uveitis patients. Uveitic activity causes fluctuating IOP due to decreased Co, increased uveoscleral outflow or decreased aqueous production.

Specific Aim 1: To evaluate the risk factors for high IOP and low Co in uveitis Hypothesis: Decreased Co and increased IOP will occur with increasing anterior chamber (AC) flare, AC cells, degree of synechial angle closure, increased duration of disease, higher uveitis activity and increasing steroid use Specific Aim 2: To determine prospectively the effect of AC flare on Co and IOP in "quiescent" uveitis Hypothesis: AC flare even in the absence of AC cells will cause progressive decline in Co.

Methods: In this proof of concept study, thirty consecutive patients with acute or chronic uveitis will be recruited from the uveitis clinic. Ten patients with "quiescent" uveitis (no AC cells) will be recruited for the prospective arm and followed every 2-3 months for 3 visits. Co will be measured using 2-minute pneumatonometer tonography. The effect of risk factors on IOP and Co in uveitis will be studied using generalized linear modelling techniques. These risk factors include AC flare (using the laser flare meter), AC cells, degree of angle closure (by gonioscopy), duration of disease, disease activity and corticosteroid use within the last year. In the prospective study, the patients will be divided into subgroups with low flare (< 20ph/ms) and high flare (≥ 20 ph/msec) and the change in Co and IOP will be analyzed.

Impact: This will be the first study to systematically analyze the risk factors for decrease in Co and increase in IOP in uveitis and to prospectively evaluate the effect of AC flare on Co. Proof that AC flare can damage the trabecular meshwork will corroborate previous experimental evidence and change the paradigm of uveitis treatment. Knowledge of the risk factors that affect Co and IOP will aid in identifying patients that may need escalation of their uveitis or glaucoma treatment to prevent optic nerve damage.

DETAILED DESCRIPTION:
Prospective subjects will be identified from the patient population pool in the Uveitis Clinic at the Truhlsen Eye Institute, University of Nebraska Medical Center, Department of Ophthalmology and Visual Sciences.

The procedures below will be performed at the first visit in all patients and at the patient's return visit in the 10 patients recruited for the prospective arm of the study (upto a maximum of 3 follow up visits)

The following information will be extracted from the chart. These are obtained routinely as part of routine clinical care through history and ocular examination by slit lamp examination and applanation tonometry for intraocular pressure measurements.

1. Age
2. Race
3. Gender
4. Diagnosis
5. Duration of disease
6. Medications, dose and duration currently and over the past year
7. Visual acuity- snellen and peripheral visual fields
8. Intraocular pressure
9. Gonioscopy: documentation of degree of synechial angle closure
10. Slit lamp examination and documentation of parameters of ocular inflammation: cells, flare, posterior synechaie extent and clock hours
11. Fundus examination

Testing done solely for the study will involve:

1. Tonographic Outflow facility: will be assessed using the pneumatonography. A two (2) minute tonography protocol will be used. The subject will be in a supine position as the weighted pneumatonometer probe is placed on the eye measuring aqueous outflow. The patient may need another drop of proparacaine prior to the test if the previous anesthesia is insufficient. This procedure should take 3-4 minutes.
2. Aqueous flare meter: The anterior chamber flare will be measured in a non-invasive way using the AC flare meter. This process will take 2-3 minutes and does not require any additional topical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years or older
2. Subjects have a diagnosis of uveitis
3. Ability to cooperate for tonography

Exclusion Criteria:

1. Any current corneal abrasion
2. Hypersensitivity to proparacaine
3. history of vitrectomy
4. hypotony (Intraocular pressure < 5 mm Hg)
5. aphakia

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective subjects will be identified from the patient population pool in the Uveitis Clinic at the Truhlsen Eye Institute, University of Nebraska Medical Center, Department of Ophthalmology and Visual Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
change in Aqeuous outflow facility | 9 months
  tonographic outflow facility calculations using pneumatonography

SECONDARY OUTCOMES:
change in intraocular pressure measured by pneumatonometer | 9 months during the study and previous 1 year historical eye pressure
  pneumatonometer measurement

CONTACTS AND LOCATIONS:
Overall Officials: Deepta Ghate, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No